CLINICAL TRIAL: NCT03391440
Title: An Open-Lable Multicenter Prospective Non-Randomized Trial to Assess the Efficacy and Safety of Morinidazole With Levofloxacin and Sequential of Levofloxacin in Women With Pelvic Inflammatory Disease
Brief Title: A Trial to Assess the Efficacy and Safety of Morinidazole in Women With Pelvic Inflammatory Disease
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HS-10090-401
Record Dates: First submitted 2017-11-28; First posted 2018-01-05 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2017-11

CONDITIONS: Pelvic Inflammatory Disease
MeSH Terms: conditions — Pelvic Inflammatory Disease | interventions — morinidazole

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- morinidazole (Experimental): morinidazole and sodium chloride injection (500 mg intravenous, twice daily for 14 days) with levofloxacin hydrochloride and sodium chloride injection (500 mg intravenous, once daily for the first week) sequential of levofloxacin hydrochloride tablets (500 mg (500 mg orally, once daily for the second week)
  Interventions: Drug: morinidazole

INTERVENTIONS:
Drug: morinidazole — morinidazole and sodium chloride injection (500 mg intravenous, twice daily for 14 days) with levofloxacin hydrochloride and sodium chloride injection (500 mg intravenous, once daily for the first week) sequential of levofloxacin hydrochloride tablets (500 mg (500 mg orally, once daily for the second week)

SUMMARY:
To assess the efficacy, safety and Population Pharmacokinetic (PPK) of morinidazole and sodium chloride injection with levofloxacin hydrochloride and sodium chloride injection sequential of levofloxacin hydrochloride tablets in women with pelvic inflammatory disease: An Open-Lable Multicenter Prospective Non-Randomized Trial

DETAILED DESCRIPTION:
Pelvic inflammatory disease (PID) is a spectrum of upper genital tract inflammations comprising endometritis, salpingitis, parametritis, oophoritis, tubo-ovarian abscess and/or pelvic peritonitis. The objectives of administering antimicrobial therapy in patients with PID are to control the symptoms and to prevent the late sequelae of the disease. Because anaerobe infections (e.g., Bacteroides fragilis infections) are associated with tubal and epithelial damage, anaerobic coverage is routinely recommended in women with pelvic infection. Guidelines have been developed in both the USA and Europe with regard to PID management. Metronidazole, a member of the nitroimidazole drug class, is included in the regimens recommended for improving anaerobic bacteria coverage. The sideeffects of metronidazole include a metallic taste, nausea, transient neutropenia, and peripheral neuropathy. Antimicrobial resistance to metronidazole has emerged after several decades of worldwide use of the drug. Morinidazole, a National Class I Antimicrobial, is a new type of third-generation nitroimidazole antimicrobial that is used for treating amoebiasis, trichomoniasis, and anaerobic bacterial infections, and which exhibits greater activity and less toxicity than metronidazole.

Morinidazole and Sodium Chloride Injection used in PID or appendicitis cases had been approved by CFDA in 2014. This phase 4 study is to assess the efficacy, safety and Population Pharmacokinetic (PPK) of morinidazole in PID.

ELIGIBILITY:
Inclusion Criteria:

* women between 18 and 65 years old
* patients with the diagnosis of PID:

  1. sexually active women or women have the risk of sexually transmitted infections, and
  2. lower abdominal pain symptoms, and
  3. lower abdominal tenderness, and adnexal and cervical motion tenderness on bimanual vaginal examination, and
  4. as well as at least one of the following signs:

     1. pyrexia (axillary temperature > 37.8 °C)
     2. mucopurulent cervical or vaginal discharge
     3. an elevated vaginal discharge white blood cell count (WBC)
     4. an elevated erythrocyte sedimentation rate
     5. an elevated C-reactive protein
     6. laboratory tests confirmed the presence of Chlamydia trachomatis infection in the cervix
     7. WBC > 10*109/L on routine blood examination
  5. Voluntary signing of written informed consent

Exclusion Criteria:

* patients with a history of antibiotic therapy for more than 3 days
* patients with any condition likely to require surgery
* Cervical / vaginal discharge examination found Gonorrhea gonorrhea
* patients with an allergy to nitroimidazole or quinolones
* patients with brain and spinal cord lesions, epilepsy and various organ sclerosis
* patients who received an abortion or surgery of uterus, cervix, abdomen within 1 month
* serious chronic liver disease (Child-Pugh graded C-class)
* patients with hematopoietic dysfunction or chronic alcoholism
* any factors that increase the risk of QTc prolongation or arrhythmia
* ALT and / or AST ≥ 2 times the ULN
* serum creatinine ≥ 1.5 times the ULN
* total bilirubin ≥ 1.5 times the ULN
* ECG QTc interval> 470ms
* any clinically significant abnormalities in rhythms, conduction or morphology of resting ECGs
* Pregnant women, breastfeeding women, women of childbearing age without effective contraceptive

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 469 (Estimated)
Dates: Start 2016-09 (Actual); Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Clinical cure Rate | 7-30 days
  Clinical cure Rate （according to symptoms and signs） at 7-30 days post-therapy

SECONDARY OUTCOMES:
The incidence of AE | 14 days
  The incidence of adverse events
Incidence of ADR | 14 days
  Incidence of adverse reactions
Incidence of serious ADR | 14 days
  Incidence of serious adverse reactions
Bacteriological response（Bacterial elimination rate） | the first day and 7-30 days
  Bacteriological response (on the first day post-therapy, at 7-30 days post-therapy)
PPK parameters | 14 days
  Area under the plasma concentration versus time curve (AUC) of morinidazole

CONTACTS AND LOCATIONS:
Locations (1):
- Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei, China